CLINICAL TRIAL: NCT03975530
Title: Piloting a Precision Approach to Home Visiting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: Inter-Tribal Council of Michigan, Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 9315
Record Dates: First submitted 2019-05-22; First posted 2019-06-05 (Actual); Last update posted 2022-01-06 (Actual); Status verified 2022-01

CONDITIONS: Parenting; Mother-Child Relations; Child Development
Keywords: Home visiting interventions; American Indian; Community based participatory research; Pregnancy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Precision Family Spirit (Experimental): Family Spirit home-visiting sites from the Inter-Tribal Council of Michigan (ITC of MI) will be selected based on comparability and randomized to provide either Standard Family Spirit or Precision Family Spirit to their clients. The investigators will select four sites and randomize two of them to Standard Family Spirit and two to Precision Family Spirit. Both groups will receive educational Family Spirit lessons. Each lesson will take about 60 minutes. Participants will receive a customized version of Family Spirit that is unique to your circumstances. The two sites randomized to provide the Precision approach will receive additional training on how to provide it. At 6 months postpartum, and upon completion of the intervention, participants in the treatment group will be asked to participate in brief semi-structured phone interviews.
  Interventions: Behavioral: Precision Family Spirit
- Standard Family Spirit (Active Comparator): Family Spirit home-visiting sites from the Inter-Tribal Council of Michigan (ITC of MI) will be selected based on comparability and randomized to provide either Standard Family Spirit or Precision Family Spirit to their clients. The investigators will select four sites and randomize two of them to Standard Family Spirit and two to Precision Family Spirit. Both groups will receive educational Family Spirit lessons. Each lesson will take about 60 minutes. Participants will receive Family Spirit lessons based on a standard program schedule.
  Interventions: Behavioral: Standard Family Spirit

INTERVENTIONS:
Behavioral: Precision Family Spirit — Family Spirit home-visiting sites from the Inter-Tribal Council of Michigan (ITC of MI) will be selected based on comparability and randomized to provide either Standard Family Spirit or Precision Family Spirit to their clients. Both groups will receive educational Family Spirit lessons. Each lesson will take about 60 minutes. Participants will receive a customized version of Family Spirit that is unique to your circumstances. The two sites randomized to provide the Precision approach will receive additional training on how to provide it.
  Arms: Precision Family Spirit
Behavioral: Standard Family Spirit — Family Spirit home-visiting sites from the Inter-Tribal Council of Michigan (ITC of MI) will be selected based on comparability and randomized to provide either Standard Family Spirit or Precision Family Spirit to their clients. The investigators will select four sites and randomize two of them to Standard Family Spirit and two to Precision Family Spirit.Both groups will receive educational Family Spirit lessons. Each lesson will take about 60 minutes. Participants will receive Family Spirit lessons based on a standard program schedule.
  Arms: Standard Family Spirit

SUMMARY:
The proposed study will be a randomized pilot study. Family Spirit home-visiting sites from the Inter-Tribal Council of Michigan (ITC of MI) will be selected based on comparability and randomized to provide either standard Family Spirit or precision Family Spirit to their clients. Sites in both groups will use an electronic platform to support implementation. The investigators will select four sites and randomize two of them to standard Family Spirit and two to precision Family Spirit. Sites will be matched based on annual volume of clients served and geographic similarity (i.e. urban vs. rural). All participating sites will be trained in the electronic implementation support platform. The two sites randomized to provide the precision approach will receive additional training on how to provide it.

In each site, all new clients who are prenatal or up to 2-months postpartum will be offered participation in the study. The study will then follow them until 12 months postpartum and measure outcomes during this time (see measurement table below). Qualitative interviews with precision participants will be done at 6 and 12 months postpartum. Focus group discussions with home visitors will also be completed during regular study team meetings. Analysis of study instruments (basic psychometrics based on baseline and end line data) and preliminary differences between the sites on Aim 3 and 4 outcomes will be done in December 2019 assuming the investigators have achieved their estimated sample size with enough retention for 6-months post enrollment. Dissemination of results will be done upon completion of the analysis.

DETAILED DESCRIPTION:
Home visiting programs provide critical support to families and young children to promote healthy development and reduce health disparities. Decades of research has yielded a robust evidence base supporting their effectiveness and impact on maternal and child outcomes. In 2010, the importance of these interventions was recognized nationally with the authorization of $1.5 billion to fund Maternal, Infant, and Early Childhood Home Visiting (MIECHV) across states and tribes. MIECHV was most recently reauthorized and funded for five years in early 2018. There are now 21 evidence-based early childhood home visiting models nationwide, all of which have evidence from multiple randomized controlled trials, favorable impacts on primary and secondary outcomes, and sustained impacts of the intervention over time.

Despite robust evidence of early childhood home-visiting effectiveness, replication and scale-up beyond the context of research has been challenging. Improving program retention, enhancing program content to address families' unique and often complex needs, and increasing fidelity have been identified as priority areas for further research. While building the evidence base for home-visiting programs, researchers necessarily took a "one-size-fits-all" approach - designing programs that are often lengthy (2-3 years long) and include standard lesson sequencing and dosing delivered in the same way to all participants. However, mothers and children do not all need the same program content or dosages. A one-size-fits-all approach fails to address maternal-child need and has led to differential outcomes across studies and populations, indicating that the promise of home-visiting to improve health has yet to be fully realized.

The need for home-visiting programs that can address maternal-child diverse and emergent needs and improve client reach and retention, while maintaining fidelity to the active ingredients of evidence-based home-visiting programs, is at the forefront of research and practice-based dialogue in the US. Recent qualitative research on high- and low-retention sites within the Nurse Family Partnership network showed that nurses in high retention sites were more collaborative with families and adapted the program to align more with families' needs compared to nurses in low retention sites. Based on these findings, Ingoldsby and colleagues used principals of motivational interviewing to provide nurses with more explicit control over the visit schedule and content to families. When they compared retention rates for nurses trained in motivational interviewing to rates for nurses trained in the standard approach, they found retention rates were significantly better when nurses had more flexibility in service delivery.

For the past several years, the Johns Hopkins Center for American Indian Health (CAIH) at Johns Hopkins University has partnered with the Annie E. Casey Foundation for formative work to develop a precision public health approach to the Family Spirit home-visiting program. Leveraging CAIH's existing evidence-based home-visiting program, Family Spirit, the goal of this project was to enhance the Family Spirit model to aid home visitors in tailoring content to meet families' specific needs and continuously monitor clients' emergent issues or improvements so that home-visiting education remains responsive, relevant, and feasible. This precision approach and corresponding implementation support have been developed. The current study will be a pilot study of the precision approach compared to the standard of care. In the standard of care, families receive regular home visits, delivered in the same sequence for up to 39 months. In the precision approach, there is a core set of lessons that every mother will get, but then additional lessons will be added based on maternal or child need. For example, if a mother is a first-time mom, they will get additional baby care lessons that are included in the standard Family Spirit curriculum but may not be relevant for moms with previous children.

ELIGIBILITY:
Inclusion Criteria:

* Prenatal or postpartum females who have a baby no older than 2 months old
* At least 14 years of age at time of conception
* Receiving Family Spirit services through ITC of MI

Exclusion Criteria:

* < 13 years old at time of conception of index pregnancy
* Index child is older than 2 months of age
* Inability to participate in full intervention or evaluation

Min Age: 14 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Study participants will be pregnant or recent postpartum females aged 14 or older at time of conception of index pregnancy who are already enrolled in Family Spirit.
Enrollment: 66 (Actual)
Dates: Start 2019-06-24 (Actual); Primary Completion 2020-12-18 (Actual); Study Completion 2020-12-18 (Actual)

PRIMARY OUTCOMES:
Acceptability of the home-visiting program from the perspective of mothers enrolled | Baseline, 2-months postpartum, 6-months postpartum, 12-months postpartum
  We will use the acceptability subscale from the Applied Mental Health Research group's Implementation Measure:
  Haroz, E. E., Bolton, P., Nguyen, A. J., Lee, C., Bogdanov, S., Bass, J., ... & Murray, L. (2019). Measuring implementation in global mental health: validation of a pragmatic implementation science measure in eastern Ukraine using an experimental vignette design. BMC health services research, 19(1), 262.
  The acceptability subscale has 17 items and is scored as an average across items with a range of 0 being lowest acceptability to 3 being highest acceptability.
Retention in the home-visiting programs | 2-months postpartum, 6-months postpartum, 12-months postpartum
  We will compare the proportion of mothers who enroll and are still enrolled at the measurement timepoint across the study arms.
Participant satisfaction | 6-months postpartum, 12-months postpartum
  We will use an adapted version of the satisfaction scale used in the final Family Spirit trial:
  Barlow A, Mullany B, Neault N, et al. Paraprofessional Delivered, Home-Visiting Intervention for American Indian Teen Mothers and Children: Three-Year Outcomes from a Randomized Controlled Trial. American Journal of Psychiatry. 2015; 172(2):154-162. doi: 10.1176/appi.ajp.2014.14030332.
  For the purposes of this study, we will focus on the seven items that aimed to measure satisfaction with the skills and competencies Family Spirit aims to instill in parents (e.g., "I learned helpful skills" or "Because of what I've learned in the program, I feel that my child is healthier"). The satisfaction items are scored 0 "Strongly Disagree" to 5 "Strongly Agree," and higher total scores correlate with higher levels of satisfaction.
Adherence | Study enrollment through study completion, an average of 1 year
  We will compare the percent of prescribed visits completed at 6- and 12-months across study arms.
Home visitor-participant relationship | 2-months postpartum, 6-months postpartum, 12-months postpartum
  We will use the shortened version of the Working Alliance Inventory (WAI). It has 12 items, and the participant and home visitor each complete their own version of the measure. Possible scores for each item on the WAI ranged from 1 "Never" to 7 "Always" and are summed for a total score. A higher score on the WAI indicates a stronger therapeutic alliance.

CONTACTS AND LOCATIONS:
Overall Officials: Emily Haroz, PhD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- Inter-Tribal Council of Michigan (ITC of MI), Sault Ste. Marie, Michigan, United States

REFERENCES:
- [Derived] Ingalls A, Rebman P, Martin L, Kushman E, Leonard A, Cisler A, Gschwind I, Brayak A, Amsler AM, Haroz EE. Towards precision home visiting: results at six months postpartum from a randomized pilot implementation trial to assess the feasibility of a precision approach to Family Spirit. BMC Pregnancy Childbirth. 2022 Sep 23;22(1):725. doi: 10.1186/s12884-022-05057-4. PMID 36151535
- [Derived] Ingalls A, Barlow A, Kushman E, Leonard A, Martin L, Team PFSS, West AL, Neault N, Haroz EE. Precision Family Spirit: a pilot randomized implementation trial of a precision home visiting approach with families in Michigan-trial rationale and study protocol. Pilot Feasibility Stud. 2021 Jan 6;7(1):8. doi: 10.1186/s40814-020-00753-4. PMID 33407939